CLINICAL TRIAL: NCT05953701
Title: InspeCKD - Secondary Data Analysis of Patients at Risk for Chronic Kidney Disease (CKD) in German Primary Care Offices to Inspect CKD Prevalence, Diagnosis Rates, Diagnostic Behaviour, Treatment Patterns and Patient Characteristics
Brief Title: Secondary Data Analysis of Patients at Risk for CKD to Inspect CKD Prevalence, Diagnosis Rates, Diagnostic Behaviour, Treatment Patterns and Patient Characteristics
Acronym: InspeCKD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00351
Record Dates: First submitted 2023-06-28; First posted 2023-07-20 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Diseases; CKD; SGLT2i
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a national secondary data analysis to determine the prevalence of diagnosed and undiagnosed CKD in German primary care offices in a patient population at high risk for the development and progression of CKD. Furthermore, it addresses the question of how CKD screening, monitoring and treatment of these patients is conducted within the German primary care setting.

DETAILED DESCRIPTION:
The study does not attempt to test any specific a priori hypothesis; it is descriptive only. Data on general patient characteristics, health insurance details, participation in disease management programs and/or family doctor-centred care, diagnoses, prescriptions, surgeries, and procedures, used billable services and laboratory test results are documented during daily routine by the physician. The data used in this setting are part of routine visits, dating back a maximum of 24 months from the date of first data transfer within the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at start of the patient´s observation period
2. Having at least one of the following diseases (based on the documented ICD-10 code):

   * Type 1 diabetes
   * Type 2 diabetes
   * Hypertension
   * Cardiovascular disease, including:

     1. Coronary and/or other atherosclerosis
     2. Myocardial infarction
     3. Heart failure
     4. Peripheral arterial disease
     5. Arrythmia
     6. Stroke
3. Having at least one year (52 weeks) of observation period

Exclusion Criteria: NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients with type 1 diabetes, type 2 diabetes and/or hypertension and/or cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 800211 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with diagnosed CKD | Dating back a maximum of 24 months from the date of first data transfer
  To assess the prevalence of diagnosed and undiagnosed CKD among all eligible patients at high risk for the development and progression of CKD
Percentage of patients with undiagnosed CKD | Dating back a maximum of 24 months from the date of first data transfer
  To assess the prevalence of diagnosed and undiagnosed CKD among all eligible patients at high risk for the development and progression of CKD
Percentage of patients with undiagnosed or diagnosed CKD | Dating back a maximum of 24 months from the date of first data transfer
  To assess the prevalence of diagnosed and undiagnosed CKD among all eligible patients at high risk for the development and progression of CKD
Percentage of patients that fulfil CKD definition according to KDIGO (Kidney Disease: Improving Global Outcomes) | Dating back a maximum of 24 months from the date of first data transfer
  To assess the prevalence of diagnosed and undiagnosed CKD among all eligible patients at high risk for the development and progression of CKD

SECONDARY OUTCOMES:
Average number of serum creatinine measurements per patient per year (52 weeks) in the study period | Dating back a maximum of 24 months from the date of first data transfer
  To evaluate the use of CKD-related laboratory diagnostics in all eligible patients
Average number of UACR measurements per patient per year (52 weeks) during the study period | Dating back a maximum of 24 months from the date of first data transfer
  To evaluate the use of CKD-related laboratory diagnostics in all eligible patients
Percentage of patients with no, one, or at least two serum creatinine measurements among all eligible patients during the study period | Dating back a maximum of 24 months from the date of first data transfer
  To evaluate the use of CKD-related laboratory diagnostics in all eligible patients
Percentage of patients with no, one, or at least two UACR measurements among all eligible patients during the study period | Dating back a maximum of 24 months from the date of first data transfer
  To evaluate the use of CKD-related laboratory diagnostics in all eligible patients
Percentage of patients who did not have serum creatinine and UACR determined at least once | Dating back a maximum of 24 months from the date of first data transfer
  To evaluate the use of CKD-related laboratory diagnostics in all eligible patients
Percentage of patients in whom both serum creatinine and UACR were determined at least once | Dating back a maximum of 24 months from the date of first data transfer
  To evaluate the use of CKD-related laboratory diagnostics in all eligible patients
Percentage of patients in whom both serum creatinine and UACR were determined at least twice | Dating back a maximum of 24 months from the date of first data transfer
  To evaluate the use of CKD-related laboratory diagnostics in all eligible patients
Percentage of patients with at least two serum creatinine measurements with an interval of at least three months among all eligible patients in the study period | Dating back a maximum of 24 months from the date of first data transfer
  To evaluate the use of CKD-related laboratory diagnostics in all eligible patients
Percentage of patients with at least two UACR measurements with an interval of at least three months among all eligible patients in the study period | Dating back a maximum of 24 months from the date of first data transfer
  To evaluate the use of CKD-related laboratory diagnostics in all eligible patients
Percentage of patients with at least two UACR and serum creatinine measurements with an interval of at least three months among all eligible patients in the study period | Dating back a maximum of 24 months from the date of first data transfer
  To evaluate the use of CKD-related laboratory diagnostics in all eligible patients
Age at index date | Dating back a maximum of 24 months from the date of first data transfer
  To describe baseline characteristics among patients with diagnosed and undiagnosed CKD at index date
Sex at index date | Dating back a maximum of 24 months from the date of first data transfer
  To describe baseline characteristics among patients with diagnosed and undiagnosed CKD at index date
BMI at index date | Dating back a maximum of 24 months from the date of first data transfer
  To describe baseline characteristics among patients with diagnosed and undiagnosed CKD at index date
Concurrent medication at index date | Dating back a maximum of 24 months from the date of first data transfer
  To describe baseline characteristics among patients with diagnosed and undiagnosed CKD at index date
Comorbidities at index date | Dating back a maximum of 24 months from the date of first data transfer
  To describe baseline characteristics among patients with diagnosed and undiagnosed CKD at index date
eGFR values at index date | Dating back a maximum of 24 months from the date of first data transfer
  To describe baseline characteristics among patients with diagnosed and undiagnosed CKD at index date
UACR values at index date | Dating back a maximum of 24 months from the date of first data transfer
  To describe baseline characteristics among patients with diagnosed and undiagnosed CKD at index date
Percentage of patients among diagnosed or undiagnosed CKD patients that are treated with either/or renin-angiotensin-system-inhibitors (ACEi, ARB), SGLT2i, statin or selective mineralocorticoid receptor antagonist at index date | Dating back a maximum of 24 months from the date of first data transfer
  To evaluate the use of medication to treat CKD among patients with diagnosed and undiagnosed CKD
Percentage of patients among diagnosed or undiagnosed CKD patients that are newly initiated with either/or renin-angiotensin-system-inhibitors (ACEi, ARB), SGLT2i, statin, selective mineralocorticoid receptor antagonist within 6 months after index date | Dating back a maximum of 24 months from the date of first data transfer
  To evaluate the use of medication to treat CKD among patients with diagnosed and undiagnosed CKD
Percentage of patients with impaired kidney function | Dating back a maximum of 24 months from the date of first data transfer
  To assess the prevalence of impaired kidney function in all eligible patients

OTHER OUTCOMES:
Percentage of patients among patients with diagnosed / undiagnosed CKD with at least one measurement of serum creatinine and UACR once per year (as recommended by KDIGO or ADA) in the study period | Dating back a maximum of 24 months from the date of first data transfer
  To assess guideline adherence and achievement of target values for the use of CKD-related laboratory diagnostics, the use of recommended CKD therapies and therapeutic target values in patients with diagnosed and undiagnosed CKD
Percentage of patients among patients with diagnosed / undiagnosed CKD that reached target values for blood pressure (as recommended by KDIGO) within 6 month (26 weeks) after index date | Dating back a maximum of 24 months from the date of first data transfer
  To assess guideline adherence and achievement of target values for the use of CKD-related laboratory diagnostics, the use of recommended CKD therapies and therapeutic target values in patients with diagnosed and undiagnosed CKD
Percentage of patients among patients with diagnosed / undiagnosed CKD with guideline adherent medication as recommended by KDIGO, ADA or DEGAM within 6 month (26 weeks) after index date | Dating back a maximum of 24 months from the date of first data transfer
  To assess guideline adherence and achievement of target values for the use of CKD-related laboratory diagnostics, the use of recommended CKD therapies and therapeutic target values in patients with diagnosed and undiagnosed CKD
Time (in weeks) from first eGFR value below 60 ml/min/1.73 m2 until the second measurement of eGFR in patients who have a reported second measurement | Dating back a maximum of 24 months from the date of first data transfer
  To assess time from first eGFR value below 60 ml/min/1.73 m2 until a second estimation is performed in all eligible patients
Time (in weeks) from first UACR value above 30 mg/g until the second measurement of UACR in patients who have a reported second measurement | Dating back a maximum of 24 months from the date of first data transfer
  To assess time from first UACR value above 30 mg/g until a second measurement of UACR is performed in all eligible patients
Time (in weeks) from first UACR value above 300 mg/g until the second measurement of UACR in patients who have a reported second measurement | Dating back a maximum of 24 months from the date of first data transfer
  To assess time from first UACR value above 300 mg/g until a second measurement of UACR is performed in all eligible patients
Time (in weeks) from first fulfilment of CKD definition to coding of ICD-10 code for CKD | Dating back a maximum of 24 months from the date of first data transfer
  To assess time from first fulfilment of CKD definition to diagnosis (by ICD-10 code) in all eligible patients
Time (in weeks) from CKD diagnosis among priorly undiagnosed patients to first prescription of RASi, SGLT2i, statin or MRA (Finerenone) | Dating back a maximum of 24 months from the date of first data transfer
  To assess time from CKD diagnosis in priorly undiagnosed patients to initiation of RASi, SGLT2i, statin or Finerenone therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Koblenz, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes indicates that AZ is accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved, AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1843R00351&attachmentIdentifier=11d1d349-a28f-4018-bd7d-242cf8ec3d9f&fileName=D1843R00351_Redacted_CSR_Synopsis.pdf&versionIdentifier=